CLINICAL TRIAL: NCT05672849
Title: Safety and Efficacy of Devices Used in Fetoscopic Neural Tube Defect Repair Cases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Michael A Belfort (Other)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Sponsor-Investigator, Michael A Belfort, Chairman and Professor, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-51509
Record Dates: First submitted 2022-11-28; First posted 2023-01-05 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Neural Tube Defects
Keywords: myelomeningocele; MMC; NTD; neural tube defect; spina bifida
MeSH Terms: conditions — Neural Tube Defects; Meningomyelocele; Spinal Dysraphism | interventions — Equipment and Supplies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Modified Devices in fetoscopic NTD repair (Experimental): Single arm study. All patients will undergo fetoscopic NTD repair with the use of the modified devices.
  Interventions: Device: Modified Surgical Instruments/Devices (Sheaths and Irrigator)

INTERVENTIONS:
Device: Modified Surgical Instruments/Devices (Sheaths and Irrigator) — Patients who choose to undergo fetoscopic surgery will be offered participation in this study. All patients will undergo a fetoscopic repair of the fetal open neural tube defect with the use of the modified devices in this study.

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of devices used in patients undergoing fetoscopic neural tube defect repair.

DETAILED DESCRIPTION:
All patients who choose to undergo fetoscopic neural tube defect repair at Texas Children's Fetal Center will be offered participation in this research study by study investigators. Description of study rationale and design and a focused interview by the study coordinator to afford potential participants a formal opportunity to examine what they have learned about the research study in the course of their evaluation and discuss how they feel about enrolling in the research study. Once the patient is deemed eligible the informed consent process will be reviewed. If patients elect to participate in the study, informed consent will be obtained, and patients provided a copy of the signed consent.

Fetoscopic Procedure: The fetoscopic open neural tube defect repair procedure will be performed with the same technique in this protocol as the investigators did in the previous protocols under this IDE (NCT02230072 and NCT03794011) in terms of exteriorization of the uterus, preparation for the fetoscopic repair and repair of the open neural tube defect. This involves release of the placode, dissection of the surrounding skin, development of myofascial flaps on either side of the defect, placement of a patch to be laid on top of the placode prior to closure of the myofascial flaps, suture of the flaps over the freed placode and patch and attempted primary closure of the defect using available skin. If necessary, the surgeons will use relaxing incisions or a skin patch to provide additional mobility to the skin to be closed over the defect. If the surgeons are unable to close the skin primarily despite best fetoscopic efforts, the option of performing/completing the repair as an open procedure exists and will be offered to the subject.

Follow-Up: The investigators will follow patients for the immediate post-procedure period (until they leave the OR).

ELIGIBILITY:
Inclusion Criteria:

* Patients who elect to undergo fetoscopic neural tube defect repair

Exclusion Criteria:

* Patients who do not elect to undergo fetoscopic neural tube defect repair

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-11-14 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events | Immediate Post-Procedure period (until the leave the OR)
  Number of adverse events associated with the investigational device
Number of device defects, malfunctions, or failures | Immediate Post-Procedure period (until the leave the OR)
  Number of device defects, malfunctions, or failures and whether the device performed as intended.

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Belfort, MD, Principal Investigator — Baylor College of Medicine and Texas Children's Hospital
Locations (1):
- Texas Childrens Hospital - Pavilion for Women, Houston, Texas, United States